CLINICAL TRIAL: NCT04640090
Title: Effectiveness of a Smartphone Wellness App to Improve Mental Well-being: A Pilot Study
Brief Title: Wellness Through Mobile Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202005219
Record Dates: First submitted 2020-11-09; First posted 2020-11-23 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Musculoskeletal Diseases; Chronic Pain; Anxiety Disorders; Depression
Keywords: Musculoskeletal disease; Chronic pain; Behavioral health; Anxiety; Depression; Mobile health; Smartphone application
MeSH Terms: conditions — Musculoskeletal Diseases; Chronic Pain; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smartphone app (Experimental): All participants in this single-arm study will receive two months of subsidized, full access to the smartphone wellness application.
  Interventions: Behavioral: Smartphone app (Wysa)

INTERVENTIONS:
Behavioral: Smartphone app (Wysa) — The commercially available smartphone application, Wysa, offers evidence-based wellness tools such as supportive listening, deep breathing techniques, guided meditation, yoga, and more. Users can communicate via text to a virtual artificial intelligence (AI) chatbot and/or a human well-being coach.

SUMMARY:
This pilot project will evaluate the potential of an affordable smartphone app to improve users' mental well-being.

DETAILED DESCRIPTION:
The goal of this pilot study is to evaluate whether a smartphone wellness application has the potential to improve anxiety and depression symptoms in people who otherwise would not have access to behavioral health care. In this pilot study, participants will include patients who present to an orthopedic specialist for chronic musculoskeletal pain and who also endorse elevated anxiety and/or depression symptoms. Patients who otherwise do not have access to adequate behavioral health resources will be eligible to enroll in the study. Through the study, participants will have two months of full access to a commercially available smartphone wellness application which offers resources such as cognitive behavioral therapy via an artificial chatbot, mindfulness and deep breathing training, and text-based access to a human well-being coach. Participants' baseline and 2-month follow-up anxiety and depression symptoms will be compared. Qualitative feedback regarding the user experience with the smartphone application will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Presentation to an orthopedic specialist at the Washington University Living Well Center for a musculoskeletal condition
* Score of 55 or higher on Patient-Reported Outcomes Measurement Information System (PROMIS) Depression and/or Anxiety measures
* Advised to consider behavioral health treatment as a component of comprehensive care for a musculoskeletal condition
* Cannot or does not wish to pursue in-person behavioral health treatment (e.g., with the center psychologist)

Exclusion Criteria:

* No access to an electronic device (such as a smartphone) to download and use the wellness app and to electronically complete follow-up self-reported health measures
* In active mental health crisis (e.g., suicidal/homicidal thoughts, psychosis) which would require an escalated level of care
* Initiating care with a behavioral health specialist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-09-14 (Actual)

PRIMARY OUTCOMES:
Mean change in anxiety symptoms | 2 months
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety scores
Mean change in depression symptoms | 2 months
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression scores

SECONDARY OUTCOMES:
Mean change in anxiety symptoms | 1 month
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety scores
Mean change in depression symptoms | 1 month
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Depression scores
Mean change in physical function symptoms | 1 month and 2 months
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function scores
Mean change in pain interference symptoms | 1 month and 2 months
  Mean longitudinal change in Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference scores
Frequency of app usage | 1 month and 2 months
  Self-reported average weekly usage of the smartphone app

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
We do not have plans to share IPD from this pilot study. Requests for IPD will be considered on a case-by-case basis.

REFERENCES:
- [Background] Sheng J, Liu S, Wang Y, Cui R, Zhang X. The Link between Depression and Chronic Pain: Neural Mechanisms in the Brain. Neural Plast. 2017;2017:9724371. doi: 10.1155/2017/9724371. Epub 2017 Jun 19. PMID 28706741
- [Background] Gureje O, Von Korff M, Simon GE, Gater R. Persistent pain and well-being: a World Health Organization Study in Primary Care. JAMA. 1998 Jul 8;280(2):147-51. doi: 10.1001/jama.280.2.147. PMID 9669787
- [Background] Dahlhamer J, Lucas J, Zelaya C, Nahin R, Mackey S, DeBar L, Kerns R, Von Korff M, Porter L, Helmick C. Prevalence of Chronic Pain and High-Impact Chronic Pain Among Adults - United States, 2016. MMWR Morb Mortal Wkly Rep. 2018 Sep 14;67(36):1001-1006. doi: 10.15585/mmwr.mm6736a2. PMID 30212442
- [Background] Ruoff GE. Depression in the patient with chronic pain. J Fam Pract. 1996 Dec;43(6 Suppl):S25-33; discussion S34. PMID 8969710
- [Background] Vranceanu AM, Beks RB, Guitton TG, Janssen SJ, Ring D. How do Orthopaedic Surgeons Address Psychological Aspects of Illness? Arch Bone Jt Surg. 2017 Jan;5(1):2-9. PMID 28271080
- [Background] Andrade LH, Alonso J, Mneimneh Z, Wells JE, Al-Hamzawi A, Borges G, Bromet E, Bruffaerts R, de Girolamo G, de Graaf R, Florescu S, Gureje O, Hinkov HR, Hu C, Huang Y, Hwang I, Jin R, Karam EG, Kovess-Masfety V, Levinson D, Matschinger H, O'Neill S, Posada-Villa J, Sagar R, Sampson NA, Sasu C, Stein DJ, Takeshima T, Viana MC, Xavier M, Kessler RC. Barriers to mental health treatment: results from the WHO World Mental Health surveys. Psychol Med. 2014 Apr;44(6):1303-17. doi: 10.1017/S0033291713001943. Epub 2013 Aug 9. PMID 23931656
- [Background] Kozloff N, Sommers BD. Insurance Coverage and Health Outcomes in Young Adults With Mental Illness Following the Affordable Care Act Dependent Coverage Expansion. J Clin Psychiatry. 2017 Jul;78(7):e821-e827. doi: 10.4088/JCP.16m11357. PMID 28703947
- [Background] Inkster B, Sarda S, Subramanian V. An Empathy-Driven, Conversational Artificial Intelligence Agent (Wysa) for Digital Mental Well-Being: Real-World Data Evaluation Mixed-Methods Study. JMIR Mhealth Uhealth. 2018 Nov 23;6(11):e12106. doi: 10.2196/12106. PMID 30470676
- [Background] Kroenke K, Yu Z, Wu J, Kean J, Monahan PO. Operating characteristics of PROMIS four-item depression and anxiety scales in primary care patients with chronic pain. Pain Med. 2014 Nov;15(11):1892-901. doi: 10.1111/pme.12537. Epub 2014 Aug 19. PMID 25138978
- [Background] Lee AC, Driban JB, Price LL, Harvey WF, Rodday AM, Wang C. Responsiveness and Minimally Important Differences for 4 Patient-Reported Outcomes Measurement Information System Short Forms: Physical Function, Pain Interference, Depression, and Anxiety in Knee Osteoarthritis. J Pain. 2017 Sep;18(9):1096-1110. doi: 10.1016/j.jpain.2017.05.001. Epub 2017 May 10. PMID 28501708
- [Background] Gambassi G. Pain and depression: the egg and the chicken story revisited. Arch Gerontol Geriatr. 2009;49 Suppl 1:103-12. doi: 10.1016/j.archger.2009.09.018. PMID 19836622
- [Background] Bair MJ, Robinson RL, Katon W, Kroenke K. Depression and pain comorbidity: a literature review. Arch Intern Med. 2003 Nov 10;163(20):2433-45. doi: 10.1001/archinte.163.20.2433. PMID 14609780
- [Background] DeVeaugh-Geiss AM, West SL, Miller WC, Sleath B, Gaynes BN, Kroenke K. The adverse effects of comorbid pain on depression outcomes in primary care patients: results from the ARTIST trial. Pain Med. 2010 May;11(5):732-41. doi: 10.1111/j.1526-4637.2010.00830.x. Epub 2010 Mar 26. PMID 20353408
- [Background] Ang DC, Bair MJ, Damush TM, Wu J, Tu W, Kroenke K. Predictors of pain outcomes in patients with chronic musculoskeletal pain co-morbid with depression: results from a randomized controlled trial. Pain Med. 2010 Apr;11(4):482-91. doi: 10.1111/j.1526-4637.2009.00759.x. Epub 2009 Dec 9. PMID 20002592
- [Background] Weil TP. Insufficient dollars and qualified personnel to meet United States mental health needs. J Nerv Ment Dis. 2015 Apr;203(4):233-40. doi: 10.1097/NMD.0000000000000271. PMID 25816044
- [Background] Foraker RE, Kite B, Kelley MM, Lai AM, Roth C, Lopetegui MA, Shoben AB, Langan M, Rutledge NL, Payne PR. EHR-based Visualization Tool: Adoption Rates, Satisfaction, and Patient Outcomes. EGEMS (Wash DC). 2015 Jun 18;3(2):1159. doi: 10.13063/2327-9214.1159. eCollection 2015. PMID 26290891
- [Background] Kretzschmar K, Tyroll H, Pavarini G, Manzini A, Singh I; NeurOx Young People's Advisory Group. Can Your Phone Be Your Therapist? Young People's Ethical Perspectives on the Use of Fully Automated Conversational Agents (Chatbots) in Mental Health Support. Biomed Inform Insights. 2019 Mar 5;11:1178222619829083. doi: 10.1177/1178222619829083. eCollection 2019. PMID 30858710
- [Background] Soons P, Denollet J. Medical psychology services in dutch general hospitals: state of the art developments and recommendations for the future. J Clin Psychol Med Settings. 2009 Jun;16(2):161-8. doi: 10.1007/s10880-009-9158-7. Epub 2009 Mar 6. PMID 19266269
- [Derived] Sinha C, Cheng AL, Kadaba M. Adherence and Engagement With a Cognitive Behavioral Therapy-Based Conversational Agent (Wysa for Chronic Pain) Among Adults With Chronic Pain: Survival Analysis. JMIR Form Res. 2022 May 23;6(5):e37302. doi: 10.2196/37302. PMID 35526201
- [Derived] Leo AJ, Schuelke MJ, Hunt DM, Metzler JP, Miller JP, Arean PA, Armbrecht MA, Cheng AL. A Digital Mental Health Intervention in an Orthopedic Setting for Patients With Symptoms of Depression and/or Anxiety: Feasibility Prospective Cohort Study. JMIR Form Res. 2022 Feb 21;6(2):e34889. doi: 10.2196/34889. PMID 35039278